CLINICAL TRIAL: NCT03662659
Title: A Randomized, Open-label, Phase II Clinical Trial of Relatlimab (Anti-LAG-3) and Nivolumab in Combination With Chemotherapy Versus Nivolumab in Combination With Chemotherapy as First-Line Treatment in Patients With Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: An Investigational Study of Immunotherapy Combinations With Chemotherapy in Patients With Gastric or Gastroesophageal Junction (GEJ) Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA224-060; 2018-001069-18 (EudraCT Number)
Record Dates: First submitted 2018-09-06; First posted 2018-09-07 (Actual); Results first posted 2022-05-09 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer; Cancer of the Stomach; Esophagogastric Junction
MeSH Terms: conditions — Stomach Neoplasms | interventions — Nivolumab; XELOX; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986213 + investigator's choice chemotherapy (Experimental): BMS-986213 + XELOX or BMS-986213 + FOLFOX or BMS-986213 + SOX
  Interventions: Biological: BMS-986213; Biological: Nivolumab; Drug: XELOX; Drug: FOLFOX; Drug: SOX
- Nivolumab + investigator's choice chemotherapy (Experimental): Nivolumab + XELOX or Nivolumab + FOLFOX or Nivolumab + SOX
  Interventions: Biological: Nivolumab; Drug: XELOX; Drug: FOLFOX; Drug: SOX

INTERVENTIONS:
Biological: BMS-986213 — Relatlimab + Nivolumab specified dose on specified days
  Arms: BMS-986213 + investigator's choice chemotherapy
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
Drug: XELOX — Oxaliplatin + capecitabine
Drug: FOLFOX — Oxaliplatin + leucovorin + fluorouracil
Drug: SOX — Oxaliplatin + tegafur/gimeracil/oteracil potassium

SUMMARY:
The purpose of this study is to determine the efficacy and safety of investigational drug relatlimab plus nivolumab in combination with chemotherapy in participants with unresectable, untreated, locally advanced or metastatic gastric or GEJ cancer.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Histologically- or cytologically-confirmed diagnosis of unresectable and either locally advanced, or metastatic gastric cancer or GEJ adenocarcinoma
* No prior treatment with systemic treatment (including HER 2 inhibitors) given as primary therapy for unresectable and either locally advanced, or metastatic GC or GEJ adenocarcinoma
* Tumor tissue must be provided for biomarker analyses

Exclusion Criteria:

* Participants with HER2 positive status
* Participants with known untreated central nervous system (CNS) metastases
* Uncontrolled or significant cardiovascular disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- United States (13):
  - Local Institution - 0049, Clovis, California
  - Local Institution - 0064, Duarte, California
  - Scripps Clinic, La Jolla, California
  - Local Institution - 0040, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Local Institution - 0041, Orange, California
  - Local Institution - 0077, Santa Monica, California
  - Local Institution - 0056, Aurora, Colorado
  - Local Institution - 0062, New Haven, Connecticut
  - Local Institution - 0050, Hackensack, New Jersey
  - Local Institution - 0054, Dallas, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - Local Institution - 0052, Seattle, Washington
- Argentina (4):
  - Local Institution - 0010, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0009, Buenos Aires, Buenos Aires F.D.
  - Local Institution - 0011, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0078, CABA
- Australia (7):
  - Local Institution - 0027, Westmead, New South Wales
  - Local Institution - 0007, Herston, Queensland
  - Local Institution - 0003, Heidelberg, Victoria
  - Local Institution - 0029, Malvern, Victoria
  - Local Institution - 0008, Shepparton, Victoria
  - Local Institution - 0005, Murdoch, Western Australia
  - Local Institution - 0028, Bedford Park
- Austria (2):
  - Local Institution - 0090, Graz
  - Local Institution - 0089, Vienna
- Belgium (2):
  - Local Institution - 0091, Brussels
  - Local Institution - 0092, Leuven
- Canada (5):
  - Local Institution - 0024, Kelowna, British Columbia
  - Local Institution - 0063, Halifax, Nova Scotia
  - Local Institution - 0070, Toronto, Ontario
  - Local Institution - 0095, Québec, Quebec
  - Local Institution - 0055, Trois-Rivières, Quebec
- Chile (4):
  - Local Institution - 0002, Rancagua, L.g.bernardoohiggins
  - Local Institution - 0001, Viña del Mar, Región de Valparaíso
  - Local Institution - 0080, Santiago, Santiago Metropolitan
  - Local Institution - 0079, Santiago
- Czechia (2):
  - Local Institution - 0031, Brno
  - Local Institution - 0030, Olomouc
- France (7):
  - Local Institution - 0047, Avignon
  - Local Institution - 0073, Besançon
  - Local Institution - 0045, Dijon
  - Local Institution - 0071, Montpellier
  - Local Institution - 0043, Paris
  - Local Institution - 0072, Paris
  - Local Institution - 0046, Rouen
- Germany (10):
  - Local Institution - 0083, Cologne
  - Local Institution - 0082, Dresden
  - Local Institution - 0017, Essen
  - Local Institution - 0081, Essen
  - Local Institution - 0014, Frankfurt
  - Local Institution - 0018, Hamburg
  - Local Institution - 0012, Hanover
  - Local Institution - 0013, Heidelberg
  - Local Institution - 0015, Mannheim
  - Local Institution - 0016, Marburg
- Italy (3):
  - Local Institution - 0020, Milan
  - IRCCS Istituto Nazionale Tumori Milano, Milan
  - Local Institution - 0021, Roma
- Norway (3):
  - Local Institution - 0088, Bergen
  - Local Institution - 0086, Oslo
  - Local Institution - 0087, Trondheim
- Local Institution - 0093, Warsaw, Poland
- Local Institution - 0067, San Juan, Puerto Rico
- Local Institution - 0038, Singapore, Singapore
- Spain (7):
  - Local Institution - 0058, Madrid, M
  - Local Institution - 0099, Badajoz
  - Local Institution - 0098, Barcelona
  - Local Institution - 0061, Barcelona
  - Local Institution - 0059, Bilbao
  - Local Institution - 0057, Madrid
  - Local Institution - 0060, Zaragoza
- United Kingdom (7):
  - Local Institution - 0075, Manchester, Greater Manchester
  - Local Institution - 0035, Nottingham, Nottinghamshire
  - Local Institution - 0032, Coventry, West Midlands
  - Local Institution - 0036, Lancaster
  - Local Institution - 0034, London
  - Local Institution - 0069, Northwood
  - Local Institution - 0033, Southampton

REFERENCES:
- [Derived] Hegewisch-Becker S, Mendez G, Chao J, Nemecek R, Feeney K, Van Cutsem E, Al-Batran SE, Mansoor W, Maisey N, Pazo Cid R, Burge M, Perez-Callejo D, Hipkin RW, Mukherjee S, Lei M, Tang H, Suryawanshi S, Kelly RJ, Tebbutt NC. First-Line Nivolumab and Relatlimab Plus Chemotherapy for Gastric or Gastroesophageal Junction Adenocarcinoma: The Phase II RELATIVITY-060 Study. J Clin Oncol. 2024 Jun 10;42(17):2080-2093. doi: 10.1200/JCO.23.01636. Epub 2024 May 9. PMID 38723227
- [Derived] Chang X, Ge X, Zhang Y, Xue X. The current management and biomarkers of immunotherapy in advanced gastric cancer. Medicine (Baltimore). 2022 May 27;101(21):e29304. doi: 10.1097/MD.0000000000029304. PMID 35623069
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 274 participants randomized and 271 treated.
Groups:
- BMS986213 + Chemotherapy: BMS986213 Q3W + Investigator Choice (IC) Chemotherapy
- Nivolumab + Chemotherapy: Nivolumab Q3W + Investigator Choice (IC) Chemotherapy
Period: Pre-treatment
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Started (Started = Randomized) | 138 | 136
Completed (Completed = Treated) | 136 | 135
Not Completed | 2 | 1
Not completed — Participant no longer met study criteria | 1 | 1
Not completed — Other reasons | 1 | 0
Period: Treatment
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Started (Started = Treated) | 136 | 135
Completed (Completed = Continuing treatment) | 0 | 1
Not Completed | 136 | 134
Not completed — Completed Treatment | 0 | 2
Not completed — Disease Progression | 85 | 97
Not completed — Study Drug Toxicity | 19 | 9
Not completed — Death | 11 | 9
Not completed — Adverse Event unrelated to Study Drug | 7 | 6
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Poor/Non-compliance | 1 | 0
Not completed — Participant no longer meets study criteria | 1 | 0
Not completed — Other reasons | 10 | 8
Not completed — Administrative reasons by sponsor | 1 | 0
Not completed — maximum clinical benefit | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy | Total
Number analyzed (Participants) | 138 | 136 | 274
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.4 (12.1) | 61.8 (11.3) | 60.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 94 | 98 | 192
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 10 | 27
  Not Hispanic or Latino | 73 | 80 | 153
  Unknown or Not Reported | 48 | 46 | 94
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 128 | 122 | 250
  Black or African American | 0 | 1 | 1
  Asian | 5 | 3 | 8
  Asian Indian | 1 | 1 | 2
  Chinese | 0 | 5 | 5
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: BICR-Assessed Objective Response Rate (ORR) in Randomized LAG-3 Positive (>=1 %) Participants
Description: The number of LAG-3 Positive (>=1%) participants with a Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR) divided by the number of randomized LAG-3 positive (>=1%) participants in each arm; recorded between randomization date and the date of objectively documented progression [per RECISIT 1.1], death due to any cause, or date of subsequent anticancer therapy, whichever occurs first.
  CR= Disappearance of all target lesions PR= At least a 30% decrease in the sum of diameters of target lesions
Time Frame: Up to 25 months
Population: All randomized LAG-3 positive (>=1%) participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 97 | 98
Percentage of Participants | 48.5 [38.2 to 58.8] | 61.2 [50.8 to 70.9]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective response rate (ORR) based on Blinded Independent Central Review (BICR) and Investigator assessments is defined as the number of participants with a Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR) divided by the number of randomized participants in each arm; recorded between randomization date and the date of objectively documented progression [per RECISIT 1.1], death due to any cause, or date of subsequent anticancer therapy, whichever occurs first.
  CR= Disappearance of all target lesions PR= At least a 30% decrease in the sum of diameters of target lesions Progression=At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization date to the date of objectively documented progression, death due to any cause, or date of subsequent anticancer therapy, whichever occurs first (Up to 63 months)
Population: All randomized LAG-3 positive (>=1%) participants, and all randomized LAG-3 negative (<1%) participants, and all randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 138 | 136
Percentage of participants
  BICR-assessed with LAG-3 expression <1%: number analyzed (Participants) | 41 | 38
  BICR-assessed with LAG-3 expression <1% | 26.8 [14.2 to 42.9] | 36.8 [21.8 to 54.0]
  BICR-assessed Overall | 27.5 [20.3 to 35.8] | 41.9 [33.5 to 50.7]
  Investigator-assessed with LAG-3 expression >=1%: number analyzed (Participants) | 97 | 98
  Investigator-assessed with LAG-3 expression >=1% | 53.6 [43.2 to 63.8] | 54.1 [43.7 to 64.2]
  Investigator-assessed with LAG-3 expression <1%: number analyzed (Participants) | 41 | 38
  Investigator-assessed with LAG-3 expression <1% | 36.6 [22.1 to 53.1] | 42.1 [26.3 to 59.2]
  Investigator-assessed Overall | 48.6 [40.0 to 57.2] | 50.7 [42.0 to 59.4]

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of Response (DOR) based on Blinded Independent Central Review (BICR) and investigator is defined as the time between the date of first documented complete response (CR) or partial response (PR) and the date of the first disease progression, per RECIST 1.1, or death due to any cause, or date of subsequent anticancer therapy, whichever occurs first.
  CR= Disappearance of all target lesions PR= At least a 30% decrease in the sum of diameters of target lesions
Time Frame: From the date of first dose to the date of the first disease progression or death due to any cause, or date of subsequent anticancer therapy, whichever occurs first (Up to 63 months)
Population: All randomized responders with LAG-3 positive (>=1%), and all randomized responders with LAG-3 negative (<1%), and all randomized responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 67 | 69
Months
  BICR-assessed with LAG-3 expression >=1%: number analyzed (Participants) | 27 | 43
  BICR-assessed with LAG-3 expression >=1% | 7.72 [4.37 to 9.95] | 10.78 [5.85 to 20.67]
  BICR-assessed with LAG-3 expression <1%: number analyzed (Participants) | 11 | 14
  BICR-assessed with LAG-3 expression <1% | 5.44 [3.06 to 7.00] | 5.55 [3.48 to 9.95]
  BICR-assessed Overall: number analyzed (Participants) | 38 | 57
  BICR-assessed Overall | 5.68 [5.32 to 9.63] | 6.93 [5.55 to 12.25]
  Investigator-assessed with LAG-3 expression >=1%: number analyzed (Participants) | 52 | 53
  Investigator-assessed with LAG-3 expression >=1% | 6.21 [4.47 to 7.82] | 10.28 [7.06 to 15.61]
  Investigator-assessed with LAG-3 expression <1%: number analyzed (Participants) | 15 | 16
  Investigator-assessed with LAG-3 expression <1% | 5.54 [3.02 to 7.43] | 8.31 [6.28 to 14.13]
  Investigator-assessed Overall | 5.88 [4.47 to 6.93] | 9.92 [7.13 to 13.60]

4. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time between the date of randomization and the date of death due to any cause. For those without documentation of death, OS will be censored on the last date the participant was known to be alive.
Time Frame: From the date of randomization to the date of death due to any cause (Up to 63 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 138 | 136
Months
  LAG-3 Expression >=1%: number analyzed (Participants) | 97 | 98
  LAG-3 Expression >=1% | 14.19 [11.89 to 18.56] | 14.98 [10.02 to 21.98]
  LAG-3 Expression <1%: number analyzed (Participants) | 41 | 38
  LAG-3 Expression <1% | 9.72 [6.64 to 12.75] | 15.51 [11.43 to 17.61]
  Overall | 12.65 [10.91 to 14.49] | 15.15 [11.50 to 17.61]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Progression-Free Survival (PFS) per Blinded Independent Central Review (BICR) and Investigator is defined as the time between the date of randomization and the first date of documented progression, or death due to any cause, or date of subsequent anticancer therapy, whichever occurs first. Participants who die without a reported prior progression (and die without start of subsequent therapy) will be considered to have progressed on the date of death.
  Progression=At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From the date of randomization to the first date of documented progression, or death due to any cause, or date of subsequent anticancer therapy, whichever occurs first (Up to 63 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 138 | 136
Months
  BICR-assessed LAG-3 Expression >=1%: number analyzed (Participants) | 97 | 98
  BICR-assessed LAG-3 Expression >=1% | 7.26 [6.64 to 11.07] | 10.84 [7.43 to 15.70]
  BICR-assessed LAG-3 Expression <1%: number analyzed (Participants) | 41 | 38
  BICR-assessed LAG-3 Expression <1% | 6.80 [5.98 to 8.80] | 10.45 [6.11 to 13.70]
  BICR-assessed Overall | 7.13 [6.74 to 9.82] | 10.45 [7.13 to 12.65]
  Investigator-assessed LAG-3 Expression >=1%: number analyzed (Participants) | 97 | 98
  Investigator-assessed LAG-3 Expression >=1% | 6.97 [5.78 to 8.34] | 8.31 [5.88 to 9.72]
  Investigator-assessed LAG-3 Expression <1%: number analyzed (Participants) | 41 | 38
  Investigator-assessed LAG-3 Expression <1% | 5.39 [4.37 to 7.98] | 9.69 [6.87 to 13.70]
  Investigator-assessed Overall | 6.64 [5.52 to 7.62] | 8.31 [6.90 to 11.04]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with any grade adverse events (AEs), serious adverse events (SAE), and adverse events leading to discontinuation using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v 5.0). An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. SAE is defined as any untoward medical occurrence that, at any dose results in death, is life threatening, requires inpatient hospitalization, results in significant disability, is a birth defect, or is an important medical event.
Time Frame: From first dose to 30 days post last dose (Up to 60 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 136 | 135
Participants
  Adverse Events (AEs) | 135 | 135
  Serious Adverse Events (SAEs) | 99 | 87
  Adverse Events leading to discontinuation | 76 | 56

7. Secondary Outcome: Number of Participants Who Died
Description: Number of participants who died in each arm.
Time Frame: Up to 60 months
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 136 | 135
Participants | 122 | 118

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants with laboratory abnormalities in specific liver tests based on US conventional units. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * ALT or AST > 3 x ULN, > 5 x ULN, > 10 x ULN and > 20 x ULN
  * Total bilirubin > 2 x ULN
  * ALP > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 1.5 x ULN
  * Concurrent (within 1 day) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
  * Concurrent (within 30 days) ALT or AST > 3 x ULN and total bilirubin > 2 x ULN
Time Frame: From first dose to 30 days post last dose (Up to 60 months)
Population: All treated participants with at least one on-treatment measurement of the corresponding laboratory parameter
Measure: Count of Participants; unit: Participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 129 | 134
Participants
  ALT or AST > 3xULN | 31 | 14
  ALT or AST > 5xULN | 12 | 5
  ALT or AST > 10xULN | 4 | 1
  ALT or AST > 20xULN | 2 | 0
  TOTAL BILIRUBIN > 2xULN | 6 | 3
  ALP > 1.5xULN | 50 | 56
  CONCURRENT ALT OR AST ELEVATION > 3xULN WITH TOTAL BILIRUBIN > 1.5xULN WITHIN ONE DAY | 5 | 2
  CONCURRENT ALT OR AST ELEVATION > 3xULN WITH TOTAL BILIRUBIN > 1.5xULN WITHIN 30 DAYS | 5 | 2
  CONCURRENT ALT OR AST ELEVATION > 3xULN WITH TOTAL BILIRUBIN > 2xULN WITHIN ONE DAY | 4 | 2
  CONCURRENT ALT OR AST ELEVATION > 3xULN WITH TOTAL BILIRUBIN > 2xULN WITHIN 30 DAYS | 4 | 2

9. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests
Description: Number of participants with laboratory abnormalities in specific thyroid tests based on US conventional units. The number of participants with the following laboratory abnormalities from on-treatment evaluations will be summarized:
  * TSH value > ULN and
  * with baseline TSH value <= ULN
  * with at least one FT3/FT4 test value < LLN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values >= LLN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test.
  * TSH < LLN and
  * with baseline TSH value >= LLN
  * with at least one FT3/FT4 test value > ULN within 2-week window after the abnormal TSH test
  * with all FT3/FT4 test values <= ULN within 2-week window after the abnormal TSH test
  * with FT3/FT4 missing within 2-week window after the abnormal TSH test
Time Frame: From first dose to 30 days post last dose (Up to 60 months)
Population: All treated participants with thyroid stimulating hormone (TSH) abnormality measurement
Measure: Count of Participants; unit: Participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 129 | 133
Participants
  TSH > ULN | 39 | 43
  TSH > ULN WITH TSH <= ULN AT BASELINE: number analyzed (Participants) | 128 | 133
  TSH > ULN WITH TSH <= ULN AT BASELINE | 35 | 33
  TSH > ULN WITH AT LEAST ONE FT3/FT4 TEST VALUE < LLN | 24 | 20
  TSH > ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 15 | 19
  TSH > ULN WITH FT3/FT4 TEST MISSING | 18 | 24
  TSH < LLN | 42 | 26
  TSH < LLN WITH TSH >= LLN AT BASELINE: number analyzed (Participants) | 128 | 133
  TSH < LLN WITH TSH >= LLN AT BASELINE | 40 | 22
  TSH < LLN WITH AT LEAST ONE FT3/FT4 TEST VALUE > ULN | 22 | 11
  TSH < LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 12 | 10
  TSH < LLN WITH FT3/FT4 TEST MISSING | 19 | 11

10. Primary Outcome: BICR-Assessed Objective Response Rate (ORR) in Randomized LAG-3 Positive (>=1 %) Participants - Extended Collection
Description: The number of LAG-3 Positive (>=1%) participants with a Best Overall Response (BOR) of confirmed Complete Response (CR) or Partial Response (PR) divided by the number of randomized LAG-3 positive (>=1%) participants in each arm; recorded between randomization date and the date of objectively documented progression [per RECISIT 1.1], death due to any cause, or date of subsequent anticancer therapy, whichever occurs first.
  CR= Disappearance of all target lesions PR= At least a 30% decrease in the sum of diameters of target lesions Progression=At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study and the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: as for outcome 2
Population: All randomized LAG-3 positive (>=1%) participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
Number analyzed (Participants) | 97 | 98
Percentage of Participants | 27.8 [19.2 to 37.9] | 43.9 [33.9 to 54.3]

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose to their study completion (up to approximately 63 months). SAEs and Other AEs were assessed from first dose up to 100 days post last dose (Up to approximately 63 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | BMS986213 + Chemotherapy | Nivolumab + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 122/138 | 118/136
Serious Adverse Events (participants affected / at risk) | 110/136 | 100/135
Other Adverse Events (participants affected / at risk) | 130/136 | 133/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BMS986213 + Chemotherapy (N=136) | Nivolumab + Chemotherapy (N=135)
Anaemia (Blood and lymphatic system disorders) | 2 | 7
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 0 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Immune-mediated hypophysitis (Endocrine disorders) | 2 | 0
Lymphocytic hypophysitis (Endocrine disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3
Ascites (Gastrointestinal disorders) | 1 | 3
Colitis (Gastrointestinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 8
Dysphagia (Gastrointestinal disorders) | 4 | 9
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 3 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 8
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 6
Obstruction gastric (Gastrointestinal disorders) | 1 | 1
Oesophageal fistula (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 2 | 0
Oesophageal pain (Gastrointestinal disorders) | 1 | 0
Oesophageal perforation (Gastrointestinal disorders) | 2 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 7
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 2
General physical health deterioration (General disorders) | 3 | 6
Influenza like illness (General disorders) | 1 | 0
Medical device pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Pyrexia (General disorders) | 12 | 7
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Contrast media reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Adrenalitis (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Cholangitis infective (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 2 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1
Febrile infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Infection (Infections and infestations) | 4 | 1
Influenza (Infections and infestations) | 0 | 2
Kidney infection (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 8
Pneumonia aspiration (Infections and infestations) | 0 | 2
Post procedural infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 2
Suspected COVID-19 (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Vascular device infection (Infections and infestations) | 1 | 2
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Abdominal wall neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 | 26
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Axonal neuropathy (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Encephalitis autoimmune (Nervous system disorders) | 2 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Device dislocation (Product Issues) | 0 | 2
Device malfunction (Product Issues) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 5 | 2
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 7
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 2
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BMS986213 + Chemotherapy (N=136) | Nivolumab + Chemotherapy (N=135)
Anaemia (Blood and lymphatic system disorders) | 41 | 32
Leukopenia (Blood and lymphatic system disorders) | 5 | 7
Neutropenia (Blood and lymphatic system disorders) | 37 | 41
Thrombocytopenia (Blood and lymphatic system disorders) | 21 | 25
Hyperthyroidism (Endocrine disorders) | 10 | 3
Hypothyroidism (Endocrine disorders) | 21 | 18
Abdominal distension (Gastrointestinal disorders) | 5 | 7
Abdominal pain (Gastrointestinal disorders) | 28 | 28
Abdominal pain upper (Gastrointestinal disorders) | 16 | 12
Constipation (Gastrointestinal disorders) | 40 | 34
Diarrhoea (Gastrointestinal disorders) | 56 | 60
Dry mouth (Gastrointestinal disorders) | 12 | 9
Dyspepsia (Gastrointestinal disorders) | 7 | 7
Dysphagia (Gastrointestinal disorders) | 22 | 15
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 70 | 79
Stomatitis (Gastrointestinal disorders) | 16 | 19
Vomiting (Gastrointestinal disorders) | 49 | 49
Asthenia (General disorders) | 16 | 21
Chills (General disorders) | 8 | 6
Fatigue (General disorders) | 72 | 70
General physical health deterioration (General disorders) | 2 | 7
Mucosal inflammation (General disorders) | 16 | 12
Non-cardiac chest pain (General disorders) | 10 | 9
Oedema peripheral (General disorders) | 17 | 18
Pyrexia (General disorders) | 33 | 19
Hypersensitivity (Immune system disorders) | 8 | 3
Oral candidiasis (Infections and infestations) | 6 | 12
Pneumonia (Infections and infestations) | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 10 | 5
Urinary tract infection (Infections and infestations) | 13 | 11
Infusion related reaction (Injury, poisoning and procedural complications) | 19 | 11
Alanine aminotransferase increased (Investigations) | 15 | 16
Aspartate aminotransferase increased (Investigations) | 18 | 16
Blood alkaline phosphatase increased (Investigations) | 10 | 7
Gamma-glutamyltransferase increased (Investigations) | 9 | 8
Neutrophil count decreased (Investigations) | 25 | 16
Platelet count decreased (Investigations) | 15 | 23
Weight decreased (Investigations) | 13 | 21
White blood cell count decreased (Investigations) | 9 | 6
Decreased appetite (Metabolism and nutrition disorders) | 48 | 46
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 10 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 15
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 9
Cold dysaesthesia (Nervous system disorders) | 4 | 8
Dizziness (Nervous system disorders) | 12 | 17
Dysgeusia (Nervous system disorders) | 15 | 16
Headache (Nervous system disorders) | 16 | 9
Neuropathy peripheral (Nervous system disorders) | 39 | 48
Paraesthesia (Nervous system disorders) | 18 | 14
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 30
Polyneuropathy (Nervous system disorders) | 9 | 8
Depression (Psychiatric disorders) | 4 | 8
Insomnia (Psychiatric disorders) | 18 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 23 | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 14 | 10
Rash (Skin and subcutaneous tissue disorders) | 26 | 24
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 | 1
Hypertension (Vascular disorders) | 8 | 15
Hypotension (Vascular disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/59/NCT03662659/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT03662659/SAP_001.pdf